CLINICAL TRIAL: NCT00959114
Title: A Phase 2a, Double-Blind, Placebo Controlled Study of the Efficacy, Safety and Tolerability of 6-weeks Treatment With ALV003 In Patients With Well-Controlled Celiac Disease
Brief Title: Safety and Efficacy of ALV003 for the Treatment of Celiac Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alvine Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALV003-0921
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-07

CONDITIONS: Celiac Disease
Keywords: Celiac Disease; Coeliac Disease; Celiac Sprue; Keliakia
MeSH Terms: conditions — Celiac Disease | interventions — ALV003

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALV003 (Experimental): ALV003 is an orally administered mixture of two recombinant proteases (cysteine endoprotease B-isoform 2 and prolyl endopeptidase) engineered to degrade gluten into non-immunogenic fragments, by targeting the glutamine and proline residues common in gluten.
  Interventions: Biological: ALV003
- Placebo comparator (Placebo Comparator): Excipients for ALV003 absent the experimental compounds
  Interventions: Biological: ALV003 placebo

INTERVENTIONS:
Biological: ALV003 — ALV003 is an orally administered mixture of two enzymes (cysteine endoprotease B-isoform 2 and prolyl endopeptidase).
  Arms: ALV003
Biological: ALV003 placebo — ALV003 is an orally administered mixture of two enzymes (cysteine endoprotease B-isoform 2 and prolyl endopeptidase).
  Arms: Placebo comparator

SUMMARY:
A phase 2a study to evaluate the safety and efficacy of ALV003 to treat celiac disease.

DETAILED DESCRIPTION:
Double-blind, placebo controlled study of the efficacy, safety and tolerability of 6-weeks treatment of ALV003 in patients with well-controlled celiac disease. Approximately 110 biopsy proven celiac disease patients will be randomized to treatment with ALV003 or placebo in a 1:1 ratio. Patients will be required to have a pre-dose and a post-treatment intestinal biopsy, and also will be required to ingest a foodstuff that contains a specified amount of gluten during the active phase of the study along with the study treatment. Patients will return to the clinic weekly for the first two weeks, then every two weeks thereafter for safety visits. Patients will return to the clinic 28 days after completion of treatment for final safety and follow-up. Safety will be closely monitored throughout the study including laboratory parameters and clinical assessment of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* History of biopsy-proven celiac disease
* Adherence to a gluten-free diet
* TG2 antibody negative
* Signed informed consent

Exclusion Criteria:

* Active dermatitis herpetiformis
* History of IgE-mediated reactions to gluten
* Use of specific medications 6 months prior to entry
* History of alcohol abuse or illicit drug use
* Current untreated or GI disease
* Positive pregnancy test
* Received any experimental drug within 14 days of randomization
* Uncontrolled chronic disease or condition
* Uncontrolled complications of celiac disease
* Any medical condition, which could adversely affect participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Efficacy: Intestinal mucosal morphology | 6 weeks
Safety: Tolerability of ALV003 | 6 weeks

SECONDARY OUTCOMES:
Efficacy: Change in intestinal intraepithelial lymphocyte numbers/phenotype | 6 weeks
Efficacy: Change in serological markers of celiac disease | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marja-Leena Lähdeaho, MD, PhD, Principal Investigator — FINN-MEDI Research; Markku Mäki, Prof, MD, PhD, Study Chair — Tampere University
Locations (1):
- FINN-MEDI Research - Clinical Trials Center, Tampere, Finland

REFERENCES:
- [Derived] Lahdeaho ML, Kaukinen K, Laurila K, Vuotikka P, Koivurova OP, Karja-Lahdensuu T, Marcantonio A, Adelman DC, Maki M. Glutenase ALV003 attenuates gluten-induced mucosal injury in patients with celiac disease. Gastroenterology. 2014 Jun;146(7):1649-58. doi: 10.1053/j.gastro.2014.02.031. Epub 2014 Feb 25. PMID 24583059